CLINICAL TRIAL: NCT05677932
Title: Bright Light Therapy for Post-COVID-19 Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joey WY Chan, Associate Professor (Clinical), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.359
Record Dates: First submitted 2023-01-06; First posted 2023-01-10 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Post COVID-19 Condition
Keywords: COVID-19; Long COVID; Fatigue
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Fatigue | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial
Who Masked: Participant
Masking Description: The subjects will be explained that the study aims to test the efficacy of two different modalities of light treatments for fatigue including white light and red light, without mentioning which one is the placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright light therapy (Experimental): 10,000lux bright light
  Interventions: Device: Bright light therapy
- Placebo group (Experimental): 50 lux dim red light
  Interventions: Device: Dim red light therapy

INTERVENTIONS:
Device: Bright light therapy — Exposure to bright light therapy for 30mins a day for two weeks
  Arms: Bright light therapy
Device: Dim red light therapy — Exposure to 50lux dim red light therapy for 30mins a day for two weeks
  Arms: Placebo group

SUMMARY:
This is a randomized placebo-controlled trial to examine the efficacy of two-week bright light therapy for patients with post-COVID-19 fatigue.

DETAILED DESCRIPTION:
This randomized placebo-controlled trial aims to evaluate the efficacy of BLT in reducing fatigue symptoms after COVID-19 infection. The second aim of the study is to explore the effects of BLT on insomnia, depression and anxiety symptoms.

Method: Each eligible participant will be randomized to either i) bright light therapy (BLT) or ii) dim red light (placebo) treatment for 30-minutes daily at their habitual wake time for a total of two weeks. Participants will be evaluated at baseline, 2nd (end of treatment), and 4th week (post-treatment 2-week) for fatigue and other symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Capable to give informed consent
* COVID-19 infection confirmed by PCR test or a Rapid Antigen Test (RAT) with onset of at least three months
* Reports new onset or exacerbation of fatigue after onset of COVID-19 and lasted for over two months
* Scoring 7 or above for the item "worst level of fatigue during the last 24 hours" in the Brief Fatigue Inventory

Exclusion Criteria:

* A current or past history of bipolar disorder, schizophrenia, neurodevelopmental disorder, organic mental disorder; intellectual disabilities or substance use disorder.
* Presence of contraindications to bright light therapy: for example, history of light induced migraine/ epilepsy; current use of photosensitizing medications; presence of eye disease: e.g. retinal blindness, severe cataract, glaucoma.
* Significant medical condition/ hearing impairment/ speech deficit leading to incapability of completing clinical interview.
* Regular shift-workers
* Trans-meridian flight in the past 3 months and during the study
* Currently receiving any structured psychotherapy
* Self-reported untreated sleep disorders (e.g. severe insomnia, obstructive sleep apnea, restless leg syndrome), psychiatric illness (e.g. depression), or medical conditions associated with fatigue (e.g. anemia, heart failure, autoimmune disorders)
* Enrolment in another clinical trial of an investigational medicinal product or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change of fatigue symptoms | at 2 weeks (at the end of treatment)
  Change in the score of the Brief Fatigue Inventory (BFI). BFI ranges from 0 to 90, higher scales indicates more severe fatigue

SECONDARY OUTCOMES:
Change of insomnia symptoms | at 2 weeks (at the end of treatment)
  The change in the score of Insomnia Severity Index (ISI), which ranges from 0-28, higher score indicates higher severity of insomnia
Change of depressive symptoms | at 2 weeks (at the end of treatment)
  The change in the score of Patient Health Questionnaire -9 item (PHQ-9), which ranges from 0-27, with higher score indicates greater severity of depressive symptoms
Change of anxiety symptoms | at 2 weeks (at the end of treatment)
  The change in the score of Generalized Anxiety Disorder 7-item (GAD-7), which ranges from 0-21, with higher score indicates greater severity of anxiety symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No